CLINICAL TRIAL: NCT00002246
Title: A Pilot Open Label, Multicenter Study to Evaluate the Role of Stavudine (d4T) in the Treatment of AIDS Dementia Complex
Brief Title: A Study to Evaluate the Use of Stavudine (d4T) to Treat AIDS Dementia Complex
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Purpose: Treatment
Other Study IDs: 244E; AI455-064
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-04

CONDITIONS: AIDS Dementia Complex; HIV Infections
Keywords: AIDS Dementia Complex; Zidovudine; Stavudine; Reverse Transcriptase Inhibitors
MeSH Terms: conditions — AIDS Dementia Complex; HIV Infections | interventions — Stavudine

INTERVENTIONS:
Drug: Stavudine

SUMMARY:
The purpose of this study is to see if adding stavudine (d4T) to anti-HIV drug regimens (with or without zidovudine, ZDV) can improve symptoms of AIDS Dementia Complex (ADC, problems involving the brain or spinal cord) in HIV-positive patients.

DETAILED DESCRIPTION:
In this open-label, multicenter, multinational study, ZDV is replaced with d4T in ZDV-containing regimens, or d4T is added to non-ZDV-containing regimens in 20 patients experiencing ADC. Patients are defined as having failed treatment if they progress by one ADC stage on the MSK (Memorial Sloan Kettering) rating scale on study (i.e., from Stage 1 to 2 or Stage 2 to 3). Patients are evaluated on a weekly basis until the dementia deterioration is confirmed to be caused by HIV-1. The effect of d4T-containing regimens is assessed for the following parameters: neurological status, survival, AIDS-defining conditions, CSF (cerebrospinal fluid) and plasma viral load, CSF and blood immunological markers, blood CD4 cell counts, and viral resistance. This study also assesses the pharmacokinetics of d4T in the CSF and in the blood.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Are at least 13 years old (need consent if under 18).
* Have AIDS Dementia Complex.
* Have been on a stable anti-HIV drug regimen for at least 8 weeks prior to study entry.
* Agree to use effective methods of birth control during the study.
* Are available for at least 16 weeks of study.

Exclusion Criteria

You will not be eligible for this study if you:

* Have ever taken d4T.
* Have a neurological (brain/spinal cord) disease, such as chronic seizures or head injury, or certain other conditions that would interfere with your ability to complete the study.
* Are pregnant or breast-feeding.
* Abuse alcohol or drugs.
* Have peripheral neuropathy or a newly diagnosed AIDS-defining infection that requires treatment at the time of study enrollment.
* Have received certain medications.
* Cannot take medications by mouth.
* Have severe diarrhea for at least 7 days in a row within 30 days prior to study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 1997-10; Primary Completion 1999-03 (Actual); Study Completion 1999-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B Brew, Study Chair
Locations (5):
- United States (3):
  - HIV Neurobehavioral Research Ctr, San Diego, California
  - AIDS ReSEARCH Alliance, West Hollywood, California
  - Mount Sinai Hosp, New York, New York
- National Centre in HIV Epidemiology and Clinical Research, Sydney, Australia
- Charing Cross and Westminster Med School, London Southwest 10, United Kingdom